CLINICAL TRIAL: NCT04147845
Title: Transepidermal Delivery of Triamcinolone Acetonide or Platelet Rich Plasma Using Either Fractional Carbon Dioxide Laser or Microneedling in Treatment of Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dalia Ibrahim Halwag, Assistant Lecturer of Dermatology, Venereology and Andrology . Principal Investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlexandriaU Derma
Record Dates: First submitted 2019-10-26; First posted 2019-11-01 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Transepidermal drug delivery; Fractional Carbon Dioxide Laser; Platelet-Rich Plasma; Microneedling; Triamcinolone acetonide
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fractional Carbon dioxide laser and triamcinolone acetonide (Experimental): Group I:Fractional Carbon dioxide laser (CO2 Laser) and triamcinolone acetonide (TrA; 10 mg/ ml) (14, 15) The ablative fractional CO2 laser is delivered to the patients' scalp. The fractional ablative method is applied immediately before the topcial medication.
  Laser treatment will be given to the affected area, and immediately after the treatment, triamcinolone solution (10 mg/ml) will be dropped on the treated area and spread evenly.
  Each patient will receive four treatments, with an interval of three weeks between the treatment sessions, for a total of 12 weeks.This will be followed by a follow up period of another 4 weeks. The patients will be given no topical treatments for the alopecia areata in between the sessions. Topical post-procedure care in the form of topical antibiotics, emollient or sunscreen may be used. Each patch will be digitally macrophotographed, and evaluated clinically and by dermoscopy at baseline and at the end of the study, for signs of hair regrowth
  Interventions: Other: Fractional Carbon Dioxide Laser; Other: Triamcinolone Acetonide
- Microneedling with Dermapen and triamcinolone acetonide (Experimental): Microneedling is performed using Dermapen. This creates pin point bleeding or mild erythema which will be considered as the end point.
  Triamcinolone acetonide in concentration of 10 mg/ml (0.1 ml containing 1 mg of triamcinolone) will be applied on each lesion twice, before and after performing microneedling.
  Each patient will receive four treatments, with an interval of three weeks between the treatment sessions, for a total of 12 weeks.This will be followed by a follow up period of another 4 weeks. The patients will be given no topical treatments for the alopecia areata in between the sessions. Topical post-procedure care in the form of topical antibiotics, emollient or sunscreen may be used. Each patch will be digitally macrophotographed, and evaluated clinically and by dermoscopy at baseline and at the end of the study, for signs of hair regrowth
  Interventions: Other: Microneedling using dermapen; Other: Triamcinolone Acetonide
- Fractional Carbon dioxide laser and Platelet-rich plasma (Experimental): The same laser parameters as group I will be used, followed by application of freshly prepared PRP. The applied PRP will be spread over the whole affected area.
  Each patient will receive four treatments, with an interval of three weeks between the treatment sessions, for a total of 12 weeks.This will be followed by a follow up period of another 4 weeks. The patients will be given no topical treatments for the alopecia areata in between the sessions. Topical post-procedure care in the form of topical antibiotics, emollient or sunscreen may be used. Each patch will be digitally macrophotographed, and evaluated clinically and by dermoscopy at baseline and at the end of the study, for signs of hair regrowth
  Interventions: Other: Fractional Carbon Dioxide Laser; Other: Platelet-rich plasma
- Microneedling with Dermapen and Platelet-rich plasma (Experimental): Microneedling using dermapen is performed as Group II. Microneedling is preceeded and followed by intermittent application of freshly prepared PRP. The applied PRP will be spread over the whole affected area and again rolled till pinpoint bleeding points are noticed.
  Each patient will receive four treatments, with an interval of three weeks between the treatment sessions, for a total of 12 weeks.This will be followed by a follow up period of another 4 weeks. The patients will be given no topical treatments for the alopecia areata in between the sessions. Topical post-procedure care in the form of topical antibiotics, emollient or sunscreen may be used. Each patch will be digitally macrophotographed, and evaluated clinically and by dermoscopy at baseline and at the end of the study, for signs of hair regrowth
  Interventions: Other: Microneedling using dermapen; Other: Platelet-rich plasma

INTERVENTIONS:
Other: Fractional Carbon Dioxide Laser — The ablative fractional CO2 laser is delivered to the patients' scalp. The fractional ablative method is applied immediately before the topcial medication.
  Laser treatment will be given to the affected area, and immediately after the treatment, the treatment solution will be dropped on the treated area and spread evenly
  Arms: Fractional Carbon dioxide laser and Platelet-rich plasma; Fractional Carbon dioxide laser and triamcinolone acetonide
Other: Microneedling using dermapen — Microneedling is performed using Dermapen. This creates pin point bleeding or mild erythema which will be considered as the end point.
  The treatment solution will be applied on each lesion twice, before and after performing microneedling.
  Arms: Microneedling with Dermapen and Platelet-rich plasma; Microneedling with Dermapen and triamcinolone acetonide
Other: Triamcinolone Acetonide — triamcinolone solution (10 mg/ml) will be dropped on the treated area and spread evenly
  Arms: Fractional Carbon dioxide laser and triamcinolone acetonide; Microneedling with Dermapen and triamcinolone acetonide
Other: Platelet-rich plasma — The applied PRP will be spread over the whole affected area
  Arms: Fractional Carbon dioxide laser and Platelet-rich plasma; Microneedling with Dermapen and Platelet-rich plasma

SUMMARY:
The aim of this study is to evaluate the use of fractional carbon dioxide laser versus microneedling in the transepidermal delivery of triamcinolone acetonide and platelet rich plasma in treatment of alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is one of the most common forms of non-scarring alopecia involving the scalp and/or body. Estimated incidence of alopecia areata is 20.9 per 100,000 person-years with a cumulative lifetime incidence of 2.1%.

The exact pathophysiology of alopecia areata remains unknown. The most widely accepted hypothesis is that alopecia areata is a T cell-mediated autoimmune condition that is most likely to occur in genetically predisposed individuals.

Although, alopecia areata is a benign condition and most patients are asymptomatic, it can cause emotional and psychosocial distress in affected individuals.

First-line therapies include intralesional corticosteroids, topical corticosteroids, minoxidil, anthralin, topical immunotherapy, prostaglandin analogues, topical retinoids bexarotene, and capsaicin. Second- and third-line treatments include topical and systemic immunomodulatory therapies such as oral and topical psoralen plus UVA radiation and photodynamic therapy.No treatment is either curative or preventive. Since no single treatment option is certain to treat alopecia areata, the need for new therapies is mounting.

Intralesional corticosteroids, most commonly triamcinolone acetonide are considered a first-line treatment method for limited disease and can be used as adjunctive therapy in extensive disease. Because triamcinolone is only emulsified temporally to the water, usually it is delivered by the painful intralesional injection.

Platelet-rich plasma (PRP) has emerged as a new treatment modality in dermatology, and preliminary evidence has suggested that it might have a beneficial role in hair growth.

Drugs applied topically have the advantage of fewer side effects, and bypassing the first-pass effect. However, transepidermal dermal drug delivery has limitations, including decreased penetration of larger and water-soluble molecules.

Several strategies have been used to improve many drug penetrations into the skin: microneedling, ultrasound, and more recently transepidermal drug delivery (TED). TED is a technique based on applying a medication following an ablative method (CO2 laser, erbium lasers or ablative radiofrequency), which create vertical channels to assist the delivery of topically applied drugs into the skin. The use of nonablative lasers as well as microneedling technique has been reported with the same purpose.

Fractional laser-assisted drug delivery of corticosteroids for resistant alopecia areata is a new concept in dermatological therapy.

Microneedle devices, such as Dermaroller and Dermapen, are minimally invasive devices that bypass the stratum corneum barrier, thus accessing the skin microcirculation and achieving systemic delivery by the transepidermal route.

Trichoscopy, hair and scalp dermoscopy, is a fast, non-invasive method useful in the diagnosis and therapeutic monitoring of scalp and hair diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with alopecia areata of either gender, diagnosed both clinically and by trichoscopy
2. Patients not responding to treatment (topical and/or systemic), used properly and regularly, for at least 3 months duration

Exclusion Criteria:

1. Alopecia areata with evidence of spontaneous hair regrowth
2. Patients having active scalp inflammation or other scalp or hair diseases
3. Pregnant and lactating women
4. Patients with any bleeding disorder or receiving anti-coagulant therapy
5. Immunocompromised patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of hair regrowth | Three months
  Each patch will be digitally macrophotographed, and evaluated clinically at baseline and at the end of the treatment sessions, for signs of hair regrowth
Dermoscopic evaluation of hair regrowth | Three months
  Each patch will be digitally macrophotographed, and evaluated by dermoscopy at baseline and at the end of the treatment sessions, for signs of hair regrowth

CONTACTS AND LOCATIONS:
Overall Officials: Khaled El Mulla, MBBCh, MS, Ph.D, Study Director — Professor of Dermatology,Venereology and Andrology, Faculty of Medicine, University of Alexandria; Eman Elmorsy, MBBCh, MS, Ph.D, Study Director — Professor of Dermatology,Venereology and Andrology, Faculty of Medicine, University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT04147845/Prot_000.pdf